CLINICAL TRIAL: NCT00683345
Title: Fatigue and IL-1 Blockade in Primary Sjøgrens Syndrome
Brief Title: Fatigue and Interleukin-1 (IL-1) Blockade in Primary Sjøgrens Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: University of Oslo (Other); University of Stavanger (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P REK NORD 60/2007; 2007-000475-41 (EudraCT Number); 17772 (Other: NSD); 07/03834-7 (Other: Norwegian Medicines Agency)
Record Dates: First submitted 2008-05-20; First posted 2008-05-23 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Fatigue; Primary Sjogren
MeSH Terms: conditions — Fatigue | interventions — Interleukin 1 Receptor Antagonist Protein; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anakinra (Active Comparator): Anakinra self-administered s.c. in a dose of 100mg daily
  Interventions: Drug: Anakinra
- Placebo (Placebo Comparator): Placebo self-adminsitered s.c in a dose 0.67ml daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anakinra — Anakinra 0.67 ml (100 mg) daily subcutaneously for 4 weeks.
  Other Names: Kineret
  Arms: Anakinra
Drug: Placebo — Saline 0.67 ml daily subcutaneously as placebo drug.
  Other Names: Saline 0.9%
  Arms: Placebo

SUMMARY:
Fatigue is a prevalent phenomenon in Primary Sjøgrens syndrome (PSS). Observations indicate that the cytokine IL-1 is of importance for this phenomenon. In this study the investigators block IL-1 by giving Anakinra (an IL-1 receptor antagonist) to patients with PSS.

DETAILED DESCRIPTION:
A double-blind, placebo-controlled, parallel study of the effect on fatigue of daily injections of Anakinra for one month.

ELIGIBILITY:
Inclusion Criteria:

* Primary Sjøgrens Syndrome according to the European-American criteria
* Age 18-80 years
* Written informed consent

Exclusion Criteria:

* Hyper- og hypothyreosis
* Malignant disease
* Parkinsons disease
* Multiple sclerosis
* Conditions or diseases where Anakinra is contraindicated
* Mental depression (BDI >13)
* Neutropenia (<1.5*10.9)
* Frequent infections
* Pregnancy, lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Fatigue as measured by Fatigue Severity Scale and a visual analogue fatigue scale | 4 weeks

SECONDARY OUTCOMES:
Inflammatory cytokines and measures of oxidative stress | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roald Omdal, PhD, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Norway

REFERENCES:
- [Derived] Norheim KB, Harboe E, Goransson LG, Omdal R. Interleukin-1 inhibition and fatigue in primary Sjogren's syndrome--a double blind, randomised clinical trial. PLoS One. 2012;7(1):e30123. doi: 10.1371/journal.pone.0030123. Epub 2012 Jan 10. PMID 22253903